CLINICAL TRIAL: NCT01196728
Title: Single-centre, Randomised, Double-blind, Placebo-controlled, Four-way Crossover Clinical Study to Investigate Safety and Tolerability and Pharmacokinetics of Single Doses of CM3.1-AC100 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CellMed AG, a subsidiary of BTG plc. (Industry)
Responsible Party: Dr. Peter Geigle, Cellmed AG
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: CellMed CM3.1-AC100/03; 2010-020895-49 (EudraCT Number)
Record Dates: First submitted 2010-09-03; First posted 2010-09-08 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2010-12

CONDITIONS: Type II Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- CM3.1-AC100 dose A (Experimental): Compound CM3.1-AC100 s.c.
  Interventions: Drug: CM3.1-AC100
- CM3.1-AC100 dose B (Experimental): Compound CM3.1-AC100 s.c.
  Interventions: Drug: CM3.1-AC100
- CM3.1-AC100 dose C (Experimental): Compound CM3.1-AC100 s.c.
  Interventions: Drug: CM3.1-AC100
- Placebo (Placebo Comparator): Placebo for compound CM3.1-AC100 s.c.
  Interventions: Drug: CM3.1-AC100

INTERVENTIONS:
Drug: CM3.1-AC100 — SAD study with single ascending subcutaneous doses

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of the Glucagon-like peptide-1 (GLP-1) peptide analogue CM3.1-AC100 after single subcutaneous (sc) doses in patients with T2DM.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent prior to any study specific procedures
2. Type 2 diabetes mellitus patient, diagnostically confirmed since at least 6 months
3. Male or female patient aged 18 to 75 years at screening, both inclusive
4. BMI >22 to ≤40 kg/m2 at screening

Exclusion Criteria:

1. Type 1 diabetes mellitus, diabetes that is a result of pancreatic injury, or secondary forms of diabetes, eg Cushings's syndrome and acromegaly
2. Fasting C-peptide < 500 pM at screening
3. Acute gastrointestinal symptoms at the time of screening and/or Day -1
4. Any clinically relevant history or the presence of cardiovascular, bronchopulmonary, gastrointestinal or neurological diseases inclusive history of chronic pancreatitis or acute pancreatitis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2010-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Safety measurements | Safety will be monitored continously and safety assessments will be made on several occasions throughout the whole study
  AEs, ECGs, BP, pulse, body temperature, laboratory variables, local tolerability including a VAS score for local pain, Present Nausea Intensity (PNI) by a nausea questionnaire and a VAS score of the Overall Nausea Index (ONI)

SECONDARY OUTCOMES:
PK samples for CM3.1-AC100 | Intense PK-sampling during the 24 hours following administration of CM3.1-AC100
  Pharmacokinetics:
  AUC, AUC0-4h, AUC0-t, Cmax, tmax, t1/2lz, λz, CL/F, Vz/F of CM3.1-AC100

CONTACTS AND LOCATIONS:
Overall Officials: Peter Geigle, Dr. med., Study Chair — CellMed AG, a subsidiary of BTG plc.
Locations (1):
- Parexel International GmbH, Berlin, State of Berlin, Germany